CLINICAL TRIAL: NCT07079553
Title: Combined Effects of Transcutaneous Electrical Diaphragmatic Stimulation With ACBT's in COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0361C
Record Dates: First submitted 2025-07-03; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: COPD
Keywords: COPD, TEDS, ACBT, transcutaneous electrical diaphragmatic stimulation, Active Cycle of Breathing Techniques.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEDS + ACBT (Experimental): Participants receive transcutaneous electrical diaphragmatic stimulation (TEDS) along with active cycle of breathing techniques (ACBTs) daily for 12 weeks.
  Interventions: Device: Transcutaneous Electrical Diaphragmatic Stimulation (TEDS); Behavioral: Active Cycle of Breathing Techniques (ACBT)
- ACBT only (Active Comparator): Participants receive only active cycle of breathing techniques (ACBTs) daily for 12 weeks.
  Interventions: Behavioral: Active Cycle of Breathing Techniques (ACBT)

INTERVENTIONS:
Device: Transcutaneous Electrical Diaphragmatic Stimulation (TEDS) — TEDS was applied using surface electrodes placed over the diaphragm region. The stimulation protocol was set at 50 Hz frequency, 300 μs pulse width, with 6 seconds of stimulation followed by 5 seconds of rest, daily for 12 weeks. It was combined with ACBT sessions.
  Other Names: Active Cycle of Breathing Techniques (ACBT)
  Arms: TEDS + ACBT
Behavioral: Active Cycle of Breathing Techniques (ACBT) — ACBT sessions included breathing control, thoracic expansion exercises, and forced expiration techniques (huffing). Sessions were performed daily for 12 weeks to aid in secretion clearance and improve lung function.

SUMMARY:
The combined effects of transcutaneous electrical diaphragmatic stimulation (TEDS) and active cycle of breathing techniques (ACBTs) in patients with chronic obstructive pulmonary disease (COPD) conducted as a randomized controlled trial at Gulab Devi Hospital, the study involved 50 participants aged 40 to 60 with mild to moderate COPD. Participants were divided into two groups, one receiving both TEDS and ACBT, and the other receiving only ACBT. Over 12 weeks, improvements in lung function, oxygen saturation, exercise capacity, and quality of life were measured using spirometry, pulse oximetry, the 6-minute walk test, and the St. George's Respiratory Questionnaire. Both groups showed significant improvement, but the group receiving ACBT alone showed a slightly higher mean rank in some outcomes. The study concludes that while both interventions are beneficial, ACBT alone may offer more consistent improvements. It recommends including respiratory muscle assessments and combining interventions with education and exercise in future research.

DETAILED DESCRIPTION:
This study investigates the effectiveness of combining transcutaneous electrical diaphragmatic stimulation (TEDS) with active cycle of breathing techniques (ACBTs) in the management of chronic obstructive pulmonary disease (COPD). COPD is a progressive respiratory condition characterized by airflow limitation, respiratory muscle weakness, and reduced quality of life. Non-pharmacological interventions like pulmonary rehabilitation, including TEDS and ACBT, have shown individual benefits in improving lung function and exercise tolerance in COPD patients. However, the combined effect of these interventions has not been extensively studied.

The research was designed as a randomized controlled trial conducted at Gulab Devi Hospital, Lahore. A total of 50 patients diagnosed with mild to moderate COPD, aged between 40 and 60 years, were recruited based on defined inclusion and exclusion criteria. Participants were randomly assigned to two groups: Group A received a combination of TEDS and ACBT, while Group B received ACBT alone. The intervention lasted for 12 weeks. TEDS was applied using specific settings-50Hz frequency, 300ms width, 6 seconds of stimulation followed by 5 seconds of rest. ACBT was administered through structured sessions involving breathing control, thoracic expansion, and forced expiratory techniques.

Outcome measures included forced expiratory volume in one second (FEV₁), forced vital capacity (FVC), FEV₁/FVC ratio, oxygen saturation (both at rest and post-exercise), six-minute walk test (6MWT) distance, and the St. George's Respiratory Questionnaire (SGRQ) for quality of life assessment. Data analysis was performed using SPSS version 25, and non-parametric tests were applied due to non-normal data distribution.

ELIGIBILITY:
Inclusion Criteria:

* COPD (Mild to Moderate)
* Age: 40-60 years of both genders
* Productive cough for more than 2 months
* Oxygen saturation without Oxygen supply > 88%

Exclusion Criteria:

* Uncontrolled hypertension
* Cardiac diseases
* Active smokers

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2025-10-28 (Estimated); Study Completion 2025-11-10 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) using Spirometry | 12 weeks
  FEV1 measures the volume of air that can be forcibly exhaled in one second. It is a key indicator of airway obstruction and lung function in COPD patients.
Forced Vital Capacity (FVC) using Spirometry | 12 weeks
  FVC measures the total amount of air that can be forcibly exhaled after taking the deepest breath possible.
FEV1/FVC Ratio using Spirometry | 12 weeks
  using Spirometry
St. George's Respiratory Questionnaire (SGRQ) | baseline and at 12 weeks post intervention
  Assesses health-related quality of life specific to respiratory diseases
6-Minute Walk Test (6MWT) | Baseline and at 12 weeks post-intervention
  Assesses functional exercise capacity.

SECONDARY OUTCOMES:
Oxygen Saturation after 6-Minute Walk Test (6MWT) via Pulse Oximetry | Baseline and at 12 weeks post-intervention
  Evaluates oxygen desaturation during physical exertion, reflecting exercise tolerance and pulmonary reserve.

CONTACTS AND LOCATIONS:
Overall Officials: Arjumand Bano, MS-CPPT, Principal Investigator — Riphah International University
Locations (1):
- Arjumand, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No